CLINICAL TRIAL: NCT06256562
Title: A Multicenter, Randomized, Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of GZR18 Injection in Chinese Obese/Overweight Patients
Brief Title: A Study of GZR18 Injection in Obese/Overweight Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GL-GLP-CH2005
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2024-08

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GZR18 (Experimental): GZR18 injection s.c.
  Interventions: Drug: GZR18
- Placebo (Placebo Comparator): Placebo injection s.c.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GZR18 — Titrated to dose 1, dose 2, dose 3 or dose 4
  Arms: GZR18
Other: Placebo — Administered the same volume as GZR18
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, placebo-controlled phase II clinical study to evaluate the efficacy, safety, tolerability, and pharmacokinetics of GZR18 injection in Chinese adult obese/overweight subjects.

ELIGIBILITY:
* Inclusion Criteria:

  1. Male or female aged 18-75 years (inclusive).
  2. Obese subjects (BMI≥28 kg/m2), Or overweight subjects (24 kg/m2≤BMI<28 kg/m2) with at least one comorbidity.
  3. Able to understand the procedures and methods in this study; willing and able to maintain a stable diet and exercise lifestyle during the research period, and willing to sign the ICF voluntarily.
* Exclusion Criteria:

  1. Limb deformities or defects affecting height and body weight measurement.
  2. Pregnant or lactating women, men or women of reproductive potential unwilling to use contraception throughout the study and for 6 months after the last dose of investigational drug.
  3. History of drug abuse within 1 year before screening, or positive results in drug abuse screening during screening or before randomization.
  4. Alcohol abuse history within 6 months prior to screening.
  5. Subjects who are known or suspected to be allergic to GLP-1 drugs or excipients.
  6. Subjects with an absolute weight change greater than 5.0% due to any reason within the 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Percent (%) change from baseline in body weight at the end of the study (W30) | 30 weeks

SECONDARY OUTCOMES:
Proportion of subjects who achieved (yes/no) body weight reduction ≥5%, 10%, 15%, 20% from baseline. | 30 weeks
Weight, waist circumference, waist-to-hip ratio (waist circumference/hip circumference), and body mass index (BMI) | 30 weeks
  Changes from baseline
Percentage (%) of weight | 33 weeks
  Change from baseline at the last safety follow-up visit (W33) after discontinuation
Glucose metabolism indicators: glycated hemoglobin A1C (HbA1c), fasting plasma glucose (FPG), fasting insulin, insulin resistance index (HOMA-IR), and islet β cell function (HOMA-β) | 30 weeks
  Changes from baseline
Cardiovascular disease risk factors: blood pressure (SBP and DBP), pulse, total cholesterol (TC), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), and triglycerides (TG) | 30 weeks
  Changes from baseline
Patient-reported weight-related quality of life scores: IWQoL-Lite-CT and SF-36 scale | 30 weeks
  Changes from baseline
Anti-drug antibodies (ADAs) for GZR18 and neutralizing antibodies (NAbs) following GZR18 Injection | 33 weeks
  Changes from baseline
AUClast, AUC0-inf, Tmax, λz, t1/2, tlag, CL/F, Vz/F, AUC%extra, MRT, Css_min, Css_max, Css_av, DF, Css_min | 30 weeks
The number of adverse events (AEs)/serious adverse events (SAEs) /AEs of special interest (AESIs) that occurred during the study. | 33 weeks
Vital signs, physical examination, 12-lead Electrocardiogram (ECG), and clinical laboratory tests (hematology, urinalysis, blood biochemistry, blood amylase, blood lipase, coagulation function, calcitonin,TSH/FT3/FT4 | 33 weeks
  Change from baseline
Subject's mental health status (assessed by using the Columbia-Suicide Severity Rating Scale and Patient Health Questionnaire (PHQ-9)) | 33 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liyuan Zhao, Ph.D, Study Director — Gan & Lee Pharmaceuticals.
Locations (1):
- Gan & Lee Pharmaceuticals Co., Ltd, Beijing, China

IPD SHARING:
Plan to Share IPD: No